CLINICAL TRIAL: NCT01766622
Title: A Pilot Study of [18F]-CP18 PET/CT Imaging in Patients With Relapsed Platinum Resistant or Refractory Epithelial Ovarian Cancer, Primary Peritoneal Cancer or Fallopian Tube Cancer Therapy Receiving Birinapant, a SMAC Mimetic Therapy
Brief Title: 18F-CP18 Imaging Studies for Cancer Treatment With Birinapant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 130036; 13-C-0036
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2013-07-24

CONDITIONS: Ovarian Neoplasms; Ovarian Cancer; Fallopian Tube Neoplasms; Fallopian Tube Cancer
Keywords: Apoptosis; Pro-Apoptotic Effects; PET Imaging; TL32711; Relapsed Platinum Resistant or Refractory Epithelial Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — CP-18 compound; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

INTERVENTIONS:
Drug: [18F]-CP18 — 7mCi, IV (in the vein) at baseline
Procedure: PET/ CT — At baseline, Within 3 days after the initial Birinapant dose, A third [18F]-CP18 PET/CT will be obtained within 3 days following cycle 2, day 15 Birinapant therapy

SUMMARY:
Background:

- 18F-CP18 is a chemical designed for use in imaging studies. It is attracted to tumor cells that are being killed by cancer treatment. Researchers want to test it in imaging studies for people who are being treated with Birinapant. Birinapant is a drug used to treat advanced ovarian, fallopian tube, or peritoneal cancers. It works kills tumor cells that have not responded to earlier treatment. 18F-CP18 may help to monitor cancer treatments with this drug.

Objectives:

- To test the effectiveness of 18F-CP18 imaging studies during cancer treatment with Birinapant.

Eligibility:

- Individuals at least 18 years of age who are taking Birinapant for ovarian, fallopian tube, or peritoneal cancer.

Design:

* Participants will have a brief physical exam. They will also answer questions about their medical history and any current medications.
* Participants will receive a dose of 18F-CP18, followed by an imaging study. The study will involve a positron emission tomography/computed tomography (PET/CT) scan. The scan will last 40 minutes.
* There will be two more PET/CT scans 1 hour and 2 hours after taking 18F-CP18. These scans will look at how the tumor cells absorb and process 18F-CP18.
* This is a scanning study only. No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
Background:

Dysregulation of apoptosis is instrumental in forming the malignant phenotype and is associated with resistance to chemotherapeutics and biological therapies. Cleaved Caspase 3 (its activated form) plays a key role in the common apoptotic pathway.

CP18 is an enzyme substrate of caspase 3. The formulation [18F]-CP18 includes PEG vector which facilitates internalization and can be non-invasively imaged using PET. Once cleaved into polar fragments by caspase 3, it become trapped within the cells.

In a phase 2 NCI clinical trial (NCI Protocol (#12C0191) CTEP 9235), Birinapant (TL32711), a SMAC (second mitochondrial derived activator of caspase) mimetic, is being evaluated in patients with relapsed platinum resistant or refractory epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer.

PET/CT imaging with [18F]-CP18 may enable the non-invasive, in vivo monitoring of this drugs pro-apoptotic effects. If a measureable effect is shown in this pilot study, further evaluation of [18F]-CP18 PET/CT s potential to monitor apoptosis may be warranted.

Primary Objective:

To determine tumor uptake and retention of [18F]-CP18 before and after treatment with a SMAC mimetic (Birinapant, TL32711), in patients with relapsed platinum resistant or refractory epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer.

Eligibility:

All subjects must meet the eligibility criteria for the phase 2 study of Birinapant (NCI Protocol (#12C0191) CTEP 9235) and be enrolled in or planning to enroll in parent therapy protocol

All subjects must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed.

Design:

This is a pilot study to assess the change in [18F]-CP18 PET tumor uptake following treatment with Birinapant, a SMAC mimetic drug, in patients with relapsed platinum resistant or refractory epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer. Subjects will undergo at least 3 [18F]-CP18 PET/CT imaging studies,one pre-therapy, one within 48 hours after receiving the initial dose of Birinapant, and a third scan within 48 hours after receiving cycle 2, day 15 dose of Birinapant and prior to the tumor biopsy on the same day. An exploration of the relationship between PET imaging parameters and clinical response and various biomarkers (as determined under the referring protocol) will also be performed. Ten patients will be enrolled on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA

Subjects with pathology proven epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer that are relapsed or refractory to prior platinum-based standard care systemic regimen, enrolled, or eligible to be enrolled in the Phase 2 NCI protocol treatment using Birinapant (NCI Protocol (#12C0191)CTEP 9235); therefore must meet the inclusion criteria for that study

Ability to provide informed consent. All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of this study before any protocol related studies are performed.

EXCLUSION CRITERIA

Known allergy to any of the formulation components of [18F]-CP18.

The subject is pregnant or nursing

Participants for whom enrollment would significantly delay (> 2 weeks) the scheduled standard of care therapy.

Participants with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results are excluded.

Participants with severe claustrophobia not relieved by oral anxiolytic medication or patients weighing >136 kg (weight limit for scanner table).

Other medical conditions deemed by the PI or associates to make the patient ineligible for protocol procedures.

It is likely that all patients in this study will be surgically sterile. If this is not the case, the patient must have a negative serum beta HCG within 24 hour prior to PET/CT or be post-menopausal for greater than or equal to 2 years

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11-30; Primary Completion 2013-07-24 (Actual); Study Completion 2013-07-24 (Actual)

PRIMARY OUTCOMES:
Tumor Uptake | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Kurdziel, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Hanahan D, Weinberg RA. The hallmarks of cancer. Cell. 2000 Jan 7;100(1):57-70. doi: 10.1016/s0092-8674(00)81683-9. No abstract available. PMID 10647931
- [Background] Green AM, Steinmetz ND. Monitoring apoptosis in real time. Cancer J. 2002 Mar-Apr;8(2):82-92. doi: 10.1097/00130404-200203000-00002. PMID 11999952
- [Background] Gyrd-Hansen M, Meier P. IAPs: from caspase inhibitors to modulators of NF-kappaB, inflammation and cancer. Nat Rev Cancer. 2010 Aug;10(8):561-74. doi: 10.1038/nrc2889. PMID 20651737